CLINICAL TRIAL: NCT00105183
Title: A Double-Blind, Placebo-Controlled, Multicenter, Dose-Ranging Study of an Anti-human-T-lymphocyte Immune Globulin (EZ-2053) in the Prophylaxis of Acute Pulmonary Allograft Rejection in Adult Recipients of Primary Pulmonary Allograft(s)
Brief Title: EZ-2053 in the Prophylaxis of Acute Pulmonary Allograft Rejection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EZ-2053-001
Record Dates: First submitted 2005-03-08; First posted 2005-03-09 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary; Idiopathic Pulmonary Fibrosis; Cystic Fibrosis; Bronchiectasis; Pulmonary Vascular Disease
Keywords: pulmonary transplantation; Pulmonary Allograft Rejection
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cystic Fibrosis; Bronchiectasis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EZ-2053 (Active Comparator): Anti-human-T-lymphocyte Immune Globulin, Rabbit (EZ-2053)
  Interventions: Biological: EZ-2053
- Placebo (Placebo Comparator): USP 0.9% sodium chloride solution
  Interventions: Biological: Placebo
- EZ-2053 5mg/kg (Active Comparator): Anti-human-T-Lymphocyte Immune Globulin, Rabbit
  Interventions: Biological: EZ-2053 5mg/kg

INTERVENTIONS:
Biological: Placebo — placebo infusion, single
  Other Names: Saline
  Arms: Placebo
Biological: EZ-2053 — single IV infusion, 9 mg/kg
  Other Names: ATG; Anti-human-T-Lymphocyte Immune Globulin, Rabbit
  Arms: EZ-2053
Biological: EZ-2053 5mg/kg — single IV infusion, 5mg/kg
  Other Names: ATG; Anti-human-T-Lymphocyte Immune Globulin, Rabbit
  Arms: EZ-2053 5mg/kg

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the study drug, known as "ATG Fresenius S," which is sometimes called "EZ-2053," to prevent a lung transplant patient's body from rejecting a transplanted lung or lungs.

DETAILED DESCRIPTION:
Patients are generally consented for the study once they go on the lung transplant waiting list and then are re-consented periodically thereafter until they undergo the lung transplant surgery. A pre-surgical assessment consisting of medical history, physical exam, ECG, chest X-Ray, and blood tests are conducted. After lung transplant surgery, patients are assessed for continued eligibility. Within 6-24 hours after the end of surgery, patients are randomized to receive one infusion of study drug or placebo through a central venous catheter. Each day for 5 days following transplant surgery, patients are monitored for transplant rejection, infections, adverse events and laboratory test changes. On post-randomization Days 14, 30, 60, 90, 180, 270 and 365, patients will be monitored for acute transplant rejection, infections and cancer, pulmonary function tests and adverse experiences. Pulmonary biopsies will be performed on post-randomization Days 30, 60, 90, 180 and 365. Blood samples will be drawn during each visit.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary single or double pulmonary allograft
* Capable of understanding the purposes and risks of the study and has given written informed consent, and agrees to comply with the study requirements
* Women of childbearing potential must have a negative serum pregnancy test within 4 days prior to randomization.

Exclusion Criteria:

* Undergoing second or living donor transplant
* Prior treatment with T-cell depleting agents within the previous 5 years for the purpose of immunosuppression
* Prior plasma exchange and/or treatment with IVIg within the past 5 years
* Pulmonary infection with pan-resistant Pseudomonas or any Burkholderia species
* Known positive blood cultures
* Donor lung ischemia time > 8 hours for first lung and > 8 hours for the second lung
* Previously received or is receiving a multi-organ transplant
* Pregnant women, nursing mothers or women of child-bearing potential who are unwilling to use reliable contraception. Effective contraception must be used BEFORE beginning study drug therapy, for the duration of the study and for 6 months following completion of the study
* Active, extra-pulmonary systemic infection requiring the prolonged or chronic use of antimicrobial agents or the presence of a chronic active hepatitis B or C
* Active liver disease (liver function tests greater than or equal to 2 times the upper limit of normal)
* Severe anemia (hemoglobin, < 6 g/dL), leukopenia (WBC < 2500/mm3), thrombocytopenia (platelet count < 80,000/mm3), polycythemia (Hct > 54% [male], Hct > 49% [female]) or clinically significant coagulopathy
* Recipient or donor is seropositive for HIV
* Previous exposure or known contraindication to administration of the study drug or to rabbit proteins
* Current malignancy or a history of malignancy (within the previous 5 years), except non-metastatic basal cell or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix that has been treated successfully
* Unstable cardiovascular disease, or a myocardial infarction within the previous 6 months
* Currently participating in another clinical trial with an investigational agent and/or is taking or has been taking an investigational agent in the 30 days prior to transplant and/or has not recovered from any reversible side effects of prior investigational drug
* Unlikely to comply with visits schedule in the protocol
* Any current history of substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elbert P Trulock III, MD, Principal Investigator — Washington University School of Medicine
Locations (19):
- United States (15):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
- The Alfred Hospital, Melbourne, Victoria, Australia
- Medical University of Vienna, Vienna, Austria
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Toronto General Hospital, Toronto

RESULTS

PARTICIPANT FLOW:
Groups:
- EZ-2053 9mg/kg: Anti-human-T-lymphocyte Immune Globulin, Rabbit (EZ-2053)
Period: Overall Study
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Started | 82 (Randomized) | 79 (Randomized) | 62 (Randomized)
Completed | 60 (Completed at least 12 months follow up) | 60 (Completed at least 12 months follow up) | 39 (Completed at least 12 months follow up)
Not Completed | 22 | 19 | 23
Not completed — Death | 19 | 13 | 15
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Physician Decision | 1 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Other reason | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg | Total
Number analyzed (Participants) | 82 | 79 | 62 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 78 | 68 | 58 | 204
  >=65 years | 4 | 11 | 4 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 27 | 99
  Male | 46 | 43 | 35 | 124
Region of Enrollment [Number; unit: participants]
  United States | 45 | 41 | 36 | 122
  Canada | 5 | 5 | 5 | 15
  Austria | 18 | 18 | 14 | 50
  Australia | 14 | 15 | 7 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Event Death, Graft Loss, Acute Rejection and/or Loss to Follow-up (Whichever Occurred First)
Time Frame: 12 months
Population: ITT. During the interim analysis the 5 mg/kg arm was dropped and it was showed that the study was insufficiently powered so the main focus of study shifted to safety endpoints. Data is based on local lung biopsy readings for efficacy failure instead of central readings
Measure: Number; unit: participants
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 82 | 79 | 62
participants | 33 | 29 | 30

2. Secondary Outcome: Number of Participants With Death or Graft Loss Post-transplant
Time Frame: 12 months
Population: ITT population
Measure: Number; unit: participants
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 82 | 79 | 62
participants | 13 | 8 | 7

3. Secondary Outcome: Number of Participants With Acute Rejection
Time Frame: 12 months
Population: ITT
Measure: Number; unit: participants
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 82 | 79 | 62
participants | 22 | 20 | 22

4. Secondary Outcome: Number of Participants With Infections and Infestations
Time Frame: 12 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 82 | 78 | 61
participants | 75 | 70 | 57

5. Secondary Outcome: Number of Participants With Severe Adverse Events
Time Frame: 12 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 82 | 78 | 61
participants | 18 | 14 | 9

6. Secondary Outcome: Pulmonary Function Tests, Total Distance Walked 6 Minute Walk Test
Time Frame: 12 months
Population: Pulmonary Function Tests (PFTs) are reported for all participants of the ITT population, who were alive at 12 months after transplantation and for whom PFT results were reported for the 12-month visit
Measure: Median (Full Range); unit: Meters
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 45 | 41 | 35
Meters | 457.0 [122.0 to 714.0] | 448.0 [278.0 to 674.2] | 427.0 [0.0 to 757.0]

7. Secondary Outcome: Pulmonary Function Test, Forced Vital Capacity
Time Frame: 12 months
Population: as for outcome 6
Measure: Median (Full Range); unit: Liters
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 66 | 64 | 49
Liters | 3.0 [1.3 to 6.2] | 2.9 [1.0 to 5.1] | 3.3 [1.0 to 5.4]

8. Secondary Outcome: Pulmonary Function Test, Forced Expiratory Volume in 1 Second
Time Frame: 12 months
Population: as for outcome 6
Measure: Median (Full Range); unit: Liters
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 66 | 64 | 50
Liters | 2.3 [0.8 to 4.9] | 2.3 [0.6 to 4.4] | 2.5 [0.8 to 5.1]

9. Secondary Outcome: Pulmonary Function Test, Forced Expiratory Flow 25-75
Time Frame: 12 months
Population: as for outcome 6
Measure: Median (Full Range); unit: Liters/second
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Number analyzed (Participants) | 66 | 64 | 50
Liters/second | 2.7 [0.3 to 7.4] | 2.2 [0.3 to 9.3] | 2.6 [0.5 to 8.0]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Total number of randomized participants is 223. The total number of randomized and treated participants is 221. Two participants (1 from EZ-2053 5mg/kg group and 1 from placebo group) were randomized but were not treated and therefore not included in the adverse event reporting.
Arm/Group | EZ-2053 9mg/kg | Placebo | EZ-2053 5mg/kg
Serious Adverse Events (participants affected / at risk) | 65/82 | 52/78 | 44/61
Other Adverse Events (participants affected / at risk) | 82/82 | 78/78 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZ-2053 9mg/kg (N=82) | Placebo (N=78) | EZ-2053 5mg/kg (N=61)
Lung transplant rejection (Immune system disorders) | 9 (9) | 11 (11) | 7 (7)
Pneumonia (Infections and infestations) | 4 (4) | 6 (6) | 6 (6)
Lung infection pseudomonal (Infections and infestations) | 4 (4) | 4 (4) | 5 (5)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Enterococcal infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Alpha hemolytic streptococcal infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nocardiosis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia Escherichia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Wound infection Staphylococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ctytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Acinetobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Actinomycotic pulmonary infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bronchopulomnary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Candida pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Corynebacterium infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infectoin (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory moniliasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatic candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neisseria infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 3 (3)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obliterative Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Necrosis of bronchioli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Reperfusion injury (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Collapse of lung (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Complications of transplanted lung (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Heparin induced thrombocytopenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Anti-erythrocyte antibody (Investigations) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vertebroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Antiviral prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bronchial anastomosis (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZ-2053 9mg/kg (N=82) | Placebo (N=78) | EZ-2053 5mg/kg (N=61)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 36 (36) | 27 (27)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 38 (38) | 35 (35) | 23 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 24 (24) | 21 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 23 (23) | 19 (19)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10) | 11 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 7 (7)
Rales (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3) | 4 (4)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 3 (3)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 2 (2)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 4 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 5 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 4 (4)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 4 (4)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Sleep apnoe syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 1 (1)
Respiratory moniliasis (Infections and infestations) | 20 (20) | 21 (21) | 20 (20)
Bronchopulmonary aspergillosis (Infections and infestations) | 13 (13) | 21 (21) | 19 (19)
Lung infection Pseudomonal (Infections and infestations) | 15 (15) | 22 (22) | 19 (19)
Staphylococcal infection (Infections and infestations) | 11 (11) | 19 (19) | 11 (11)
Pneumonia (Infections and infestations) | 9 (9) | 12 (12) | 9 (9)
Cytomegalovirus viraemia (Infections and infestations) | 10 (10) | 7 (7) | 9 (9)
Cytomegalovirus infection (Infections and infestations) | 12 (12) | 8 (8) | 8 (8)
Enterococcal infection (Infections and infestations) | 10 (10) | 4 (4) | 5 (5)
Stenotrophomonas infection (Infections and infestations) | 6 (6) | 7 (7) | 7 (7)
Oral Candidiasis (Infections and infestations) | 8 (8) | 4 (4) | 2 (2)
Aspergillosis (Infections and infestations) | 3 (3) | 7 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3) | 5 (5)
Respiratory tract infection fungal (Infections and infestations) | 4 (4) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 4 (4) | 6 (6) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 6 (6) | 4 (4)
Alpha haemolytic Streptococcal infection (Infections and infestations) | 6 (6) | 4 (4) | 3 (3)
Enterobacter infection (Infections and infestations) | 6 (6) | 4 (4) | 4 (4)
Bacterial infection (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Lung infection (Infections and infestations) | 4 (4) | 5 (5) | 4 (4)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Pseudomonas infection (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Klebsiella infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 32 (32) | 46 (46) | 20 (20)
Nausea (Gastrointestinal disorders) | 44 (44) | 45 (45) | 30 (30)
Constipation (Gastrointestinal disorders) | 25 (25) | 35 (35) | 19 (19)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 12 (12) | 14 (14)
Vomiting (Gastrointestinal disorders) | 11 (11) | 16 (16) | 10 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 8 (8) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 9 (9) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 8 (8) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2) | 7 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (3) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 6 (6) | 4 (4)
Gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 5 (5) | 5 (5) | 4 (4)
Oedema peripheral (General disorders) | 39 (39) | 33 (33) | 29 (29)
Pyrexia (General disorders) | 27 (27) | 23 (23) | 15 (15)
Oedema (General disorders) | 14 (14) | 11 (11) | 13 (13)
Chest pain (Gastrointestinal disorders) | 9 (9) | 16 (16) | 7 (7)
Fatigue (General disorders) | 14 (14) | 8 (8) | 6 (6)
Asthenia (General disorders) | 7 (7) | 13 (13) | 6 (6)
Pain (General disorders) | 7 (7) | 11 (11) | 9 (9)
Chills (General disorders) | 11 (11) | 3 (3) | 7 (7)
Chest discomfort (Gastrointestinal disorders) | 5 (5) | 6 (6) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 4 (4) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 48 (48) | 42 (42) | 27 (27)
Thrombocytopenia (Blood and lymphatic system disorders) | 34 (34) | 10 (10) | 17 (17)
Leukopenia (Blood and lymphatic system disorders) | 21 (21) | 21 (21) | 14 (14)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 12 (12) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 8 (8)
Hepatic enzyme increased (Investigations) | 14 (14) | 10 (10) | 14 (14)
White blood cell count increased (Investigations) | 12 (12) | 14 (14) | 6 (6)
Blood albumin decreased (Investigations) | 7 (7) | 12 (12) | 2 (2)
Blood creatinine increased (Investigations) | 10 (10) | 9 (9) | 5 (5)
Blood urea increased (Investigations) | 3 (3) | 8 (8) | 2 (2)
Platelet count increased (Investigations) | 5 (5) | 8 (8) | 1 (1)
Blood glucose fluctuation (Investigations) | 8 (8) | 7 (7) | 5 (5)
Liver function test abnormal (Investigations) | 8 (8) | 5 (5) | 4 (4)
Platelet count decreased (Investigations) | 8 (8) | 6 (6) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3) | 7 (7) | 2 (2)
Body temperature increased (Investigations) | 7 (7) | 5 (5) | 3 (3)
Blood magnesium decreased (Investigations) | 6 (6) | 2 (2) | 5 (5)
Oxygen saturation decreased (Investigations) | 3 (3) | 6 (6) | 1 (1)
Breath sounds abnormal (Investigations) | 6 (6) | 3 (3) | 4 (4)
Troponin increased (Investigations) | 4 (4) | 2 (2) | 4 (4)
Cardiac murmur (Investigations) | 4 (4) | 5 (5) | 3 (3)
Blood uric acid increased (Investigations) | 5 (5) | 4 (4) | 1 (1)
Pulmonary function test decreased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (21) | 16 (16) | 10 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 16 (16) | 16 (16) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 12 (12) | 10 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9) | 12 (12) | 9 (9)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 10 (10) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 7 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 7 (7) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 8 (8) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 8 (8) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 26 (26) | 25 (25) | 23 (23)
Hypertension (Vascular disorders) | 26 (26) | 25 (25) | 21 (21)
Haemodynamic instability (Vascular disorders) | 9 (9) | 9 (9) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 7 (7) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 5 (5) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 23 (23) | 26 (26) | 11 (11)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 12 (12) | 7 (7)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0)
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 26 (26) | 23 (23) | 15 (15)
Tremor (Nervous system disorders) | 20 (20) | 14 (14) | 17 (17)
Dizziness (Nervous system disorders) | 16 (16) | 14 (14) | 13 (13)
Paraesthesia (Nervous system disorders) | 4 (4) | 9 (9) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 3 (3) | 4 (4)
Lethargy (Nervous system disorders) | 2 (2) | 5 (5) | 3 (3)
Somnolence (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 22 (22) | 20 (20) | 15 (15)
Tachycardia (Cardiac disorders) | 16 (16) | 16 (16) | 8 (8)
Supraventricular tachycardia (Cardiac disorders) | 7 (7) | 2 (2) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 5 (5) | 5 (5) | 4 (4)
Bradycardia (Cardiac disorders) | 5 (5) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 14 (14) | 18 (18) | 11 (11)
Insomnia (Psychiatric disorders) | 14 (14) | 18 (18) | 12 (12)
Depression (Psychiatric disorders) | 10 (10) | 11 (11) | 4 (4)
Agitation (Psychiatric disorders) | 5 (5) | 8 (8) | 3 (3)
Hallucination (Psychiatric disorders) | 8 (8) | 5 (5) | 3 (3)
Confusional state (Psychiatric disorders) | 4 (4) | 7 (7) | 3 (3)
Delirium (Psychiatric disorders) | 4 (4) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 13 (13) | 12 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (8) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (10) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 2 (2)
Renal failure (Renal and urinary disorders) | 15 (15) | 10 (10) | 16 (16)
Renal failure acute (Renal and urinary disorders) | 8 (8) | 8 (8) | 9 (9)
Renal failure chronic (Renal and urinary disorders) | 6 (6) | 6 (6) | 6 (6)
Urinary retention (Renal and urinary disorders) | 0 (0) | 3 (3) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 2 (2)
Nocturia (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (4) | 4 (4) | 2 (2)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 10 (10) | 7 (7) | 7 (7)
Pruritis (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0)
Lung transplant rejection (Immune system disorders) | 28 (28) | 33 (33) | 27 (27)
Cytokine release syndrome (Immune system disorders) | 9 (9) | 0 (0) | 6 (6)
Vision blurred (Eye disorders) | 2 (2) | 6 (6) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 5 (5) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 (6) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Interim analysis: Dropped 5mg/kg arm. Study was insufficiently powered & focus shifted to safety endpoints. Eliminated some secondary endpoints eg. steroid resistant&antibody treated rejection,CNI&antiproliferative agent, bronchiolitis obliterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protocol: The 1st publication of study results shall be a complete, joint multicenter publication or disclosure coordinated by sponsor. Later publications will reference 1st publication.

Prior to submitting for publication, the Investigator shall allow sponsor at least 30 days to review the proposed Publication. Proposed Publications shall not include either Fresenius Biotech confidential information other than the study results or personal data on any patient, such as name or initials.